CLINICAL TRIAL: NCT02546765
Title: Dexmedetomidine and IV Acetaminophen for the Prevention of Postoperative Delirium Following Cardiac Surgery in Adult Patients 60 Years of Age and Older
Brief Title: Dexmedetomidine and IV Acetaminophen for the Prevention of Postoperative Delirium Following Cardiac Surgery
Acronym: DEXACET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Balachundhar Subramaniam, Anesthesiologist, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014P000413
Record Dates: First submitted 2015-01-13; First posted 2015-09-11 (Estimated); Results first posted 2020-01-07 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Delirium
Keywords: analgesics; cardiac surgery; sedation
MeSH Terms: conditions — Delirium | interventions — Acetaminophen; Propofol; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- IV acetaminophen & IV propofol (Experimental): 20-100 µg/kg/min IV propofol given for 4-6 hours before the patients are woken up in the ICU
  1g IV acetaminophen every 6 hours for 48 hours during the first 2 days postoperatively
  Interventions: Drug: IV acetaminophen & IV propofol
- IV acetaminophen & IV dexmedetomidine (Experimental): A loading infusion of 0.5 - 1 µg/kg given over 10 minutes will be administered. After the loading infusion, a maintenance infusion of 0.1-1.4 µg/kg/hr will be initiated.
  1 g IV acetaminophen every 6 hours for 48 hours during the first 2 days postoperatively
  Interventions: Drug: IV acetaminophen & IV dexmedetomidine
- IV propofol & placebo (Active Comparator): 20-100 µg/kg/min IV propofol given for 4-6 hours before the patients are woken up in the ICU Volume of the placebo (saline) will match that of IV acetaminophen at 100ml 0.9% NaCl.
  Interventions: Drug: IV propofol & placebo
- IV dexmedetomidine & placebo (Active Comparator): 0.1-1.0 µg/kg/hour IV dexmedetomidine given for 4-6 hours before the patients are woken up in the ICU Volume of the placebo (saline) will match that of i.v. acetaminophen at 100ml 0.9% NaCl.
  Interventions: Drug: IV dexmedetomidine & placebo

INTERVENTIONS:
Drug: IV acetaminophen & IV propofol — use of IV tylenol and IV propofol for pain and sedation (respectively)
  Other Names: Ofirmev; Diprivan
  Arms: IV acetaminophen & IV propofol
Drug: IV acetaminophen & IV dexmedetomidine — use of IV tylenol and IV dexmedetomidine for pain and sedation (respectively)
  Other Names: Ofirmev; Precedex
  Arms: IV acetaminophen & IV dexmedetomidine
Drug: IV propofol & placebo — use of IV propofol for sedation and morphine, the drug of choice for cardiac pain
  Other Names: Diprivan
  Arms: IV propofol & placebo
Drug: IV dexmedetomidine & placebo — use of IV dexmedetomidine for sedation and morphine, the drug of choice for cardiac pain
  Other Names: Precedex
  Arms: IV dexmedetomidine & placebo

SUMMARY:
Investigators will assess the incidence and duration of postoperative delirium in patients ≥60 years old undergoing coronary artery bypass grafting (CABG), with/without valve surgery (aortic and/or mitral) based on different regimens for postoperative sedation and analgesia. Patients will receive either intravenous (IV) dexmedetomidine and IV acetaminophen or standard postoperative management using IV propofol with morphine or hydromorphone. The Confusion Assessment Method (CAM) will be used to assess delirium in these patients. Investigators also seek to compare postoperative (48 hours) analgesic requirements in patients with or without IV acetaminophen. Investigators will finally assess postoperative cognition in post-surgical patients up to one year post-discharge using a cognitive assessment scale.

DETAILED DESCRIPTION:
This is a prospective, randomized, placebo-controlled, triple-blinded, factorial design study consisting of 120 patients who were randomized and received a study intervention. Intravenous dexmedetomidine and acetaminophen will be compared to the standard sedation/analgesic propofol and opioid regimen.

After obtaining informed consent, study subjects will be randomized by an unblinded investigator and receive a specific combination of both sedatives and analgesic medications. Sedatives will include either IV propofol or IV dexmedetomidine, and analgesics IV acetaminophen or placebo (100 mL 0.9% NaCl equivalent to the administered volume of IV acetaminophen). Subjects will be allocated in a 1:1:1:1 fashion into the following four treatment arms: 1. IV acetaminophen with IV propofol, 2. IV acetaminophen with IV dexmedetomidine, 3. IV propofol with placebo, or 4. IV dexmedetomidine with placebo. Sedation and analgesia protocols will begin while patients are in the OR and continue as they are transferred to the Cardiovascular Intensive Care Unit (CVICU). The medications for sedation will be weight based (loading infusion of 0.5 - 1 µg/kg given over 10 minutes followed by a maintenance infusion of 0.1-1.4 µg/kg/hr for IV dexmedetomidine, or 20-100 µg/kg/min for IV propofol). Postoperative sedation is administrated 4-6 hours before patients are woken up in the CVICU. IV Acetaminophen (1g or 100mL) will be given every 6 hours for 48 hours to patients randomized to this drug. The volume of the placebo will be administered in respective groups in the same timeframe. Oral acetaminophen will be continued until discharge in all patients. All groups will also receive bolus doses of opioids (IV morphine or hydromorphone) as needed for breakthrough pain.

Patients will be administered a preoperative (baseline) and a series of post-operative evaluations to assess delirium by a blinded investigator. Baseline assessments will include the Montreal Cognitive Assessment (MoCA), days of the week (DOW), months of the year (MOY), Delirium Symptom Interview (DSI), the Geriatric Depression Scale (GDS) and the Confusion Assessment Method (CAM). Daily cognitive assessments will include the DSI, CAM, and a standard cognitive assessment. At discharge, the MoCA, DOW, MOY, DSI, and CAM will be given. Follow-up assessments will be conducted at 1 month and 1 year post-discharge and will include the telephonic MoCA, DSI, GDS and CAM. The delirium research assessments will not be provided to the treating clinicians. Treating clinicians will assess and treat delirium as usual, including assessment and correction of reversible causes, behavioral management, and use of IV haloperidol as needed for agitation. Rescue doses of haloperidol will be recorded in the study.

Blood will be collected from all subjects at the time of the baseline assessment, post-operation day 1 (POD1) while in ICU, POD 2 in the ICU, and within 48 hours of discharge. Two sets of 10 mL will be collected at each time point, with a total of 80mL of blood per patient. Efforts will be made to efficiently draw blood through the patient's arterial line at baseline or add onto to scheduled draws with phlebotomy. The plasma and buffy coat will be separated from the blood, aliquoted into labeled vials, and stored in a biomarker bank at -80°C for future use.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 60 years of age
* Undergoing CABG with/without valve (aortic and/or mitral) procedure requiring bypass

Exclusion Criteria:

* Pre-operative Left Ventricular Ejection Fraction (LVEF) < 30%
* Emergent or urgent procedures, aortic surgery
* Pre-existing cognitive impairment (defined based on a short screening assessment), Parkinson's disease, Alzheimer's disease, recent seizures (<3 months)
* Prophylactic medications for cognitive decline
* Serum creatinine > 2 mg/dl
* Liver dysfunction (liver enzymes > 4x the baseline, since patients will have a baseline liver function tests), history and exam suggestive of jaundice
* Known history of alcohol or drug abuse (>10 drinks per week)
* Hypersensitivity to any of the study drug and percutaneous procedures
* Non-English speaking

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2019-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Balachundhar Subramaniam, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Rudolph JL, Jones RN, Levkoff SE, Rockett C, Inouye SK, Sellke FW, Khuri SF, Lipsitz LA, Ramlawi B, Levitsky S, Marcantonio ER. Derivation and validation of a preoperative prediction rule for delirium after cardiac surgery. Circulation. 2009 Jan 20;119(2):229-36. doi: 10.1161/CIRCULATIONAHA.108.795260. Epub 2008 Dec 31. PMID 19118253
- [Background] Inouye SK. Delirium in older persons. N Engl J Med. 2006 Mar 16;354(11):1157-65. doi: 10.1056/NEJMra052321. No abstract available. PMID 16540616
- [Background] Saczynski JS, Marcantonio ER, Quach L, Fong TG, Gross A, Inouye SK, Jones RN. Cognitive trajectories after postoperative delirium. N Engl J Med. 2012 Jul 5;367(1):30-9. doi: 10.1056/NEJMoa1112923. PMID 22762316
- [Background] Lin YY, He B, Chen J, Wang ZN. Can dexmedetomidine be a safe and efficacious sedative agent in post-cardiac surgery patients? a meta-analysis. Crit Care. 2012 Sep 27;16(5):R169. doi: 10.1186/cc11646. PMID 23016926
- [Background] Corbett SM, Rebuck JA, Greene CM, Callas PW, Neale BW, Healey MA, Leavitt BJ. Dexmedetomidine does not improve patient satisfaction when compared with propofol during mechanical ventilation. Crit Care Med. 2005 May;33(5):940-5. doi: 10.1097/01.ccm.0000162565.18193.e5. PMID 15891317
- [Background] Shehabi Y, Grant P, Wolfenden H, Hammond N, Bass F, Campbell M, Chen J. Prevalence of delirium with dexmedetomidine compared with morphine based therapy after cardiac surgery: a randomized controlled trial (DEXmedetomidine COmpared to Morphine-DEXCOM Study). Anesthesiology. 2009 Nov;111(5):1075-84. doi: 10.1097/ALN.0b013e3181b6a783. PMID 19786862
- [Background] Maldonado JR, Wysong A, van der Starre PJ, Block T, Miller C, Reitz BA. Dexmedetomidine and the reduction of postoperative delirium after cardiac surgery. Psychosomatics. 2009 May-Jun;50(3):206-17. doi: 10.1176/appi.psy.50.3.206. PMID 19567759
- [Background] Dasta JF, Jacobi J, Sesti AM, McLaughlin TP. Addition of dexmedetomidine to standard sedation regimens after cardiac surgery: an outcomes analysis. Pharmacotherapy. 2006 Jun;26(6):798-805. doi: 10.1592/phco.26.6.798. PMID 16716133
- [Background] Holmer Pettersson P, Jakobsson J, Owall A. Plasma concentrations following repeated rectal or intravenous administration of paracetamol after heart surgery. Acta Anaesthesiol Scand. 2006 Jul;50(6):673-7. doi: 10.1111/j.1399-6576.2006.01043.x. PMID 16987360
- [Derived] Wiredu K, Mueller A, McKay TB, Behera A, Shaefi S, Akeju O. Sex Differences in the Incidence of Postoperative Delirium after Cardiac Surgery: A Pooled Analyses of Clinical Trials. Anesthesiology. 2023 Oct 1;139(4):540-542. doi: 10.1097/ALN.0000000000004656. No abstract available. PMID 37535937
- [Derived] Goncalves M, Khera T, Otu HH, Narayanan S, Dillon ST, Shanker A, Gu X, Jung Y, Ngo LH, Marcantonio ER, Libermann TA, Subramaniam B. Multivariable model of postoperative delirium in cardiac surgery patients: proteomic and demographic contributions. medRxiv [Preprint]. 2023 Oct 13:2023.05.30.23289741. doi: 10.1101/2023.05.30.23289741. PMID 37333093
- [Derived] Subramaniam B, Shankar P, Shaefi S, Mueller A, O'Gara B, Banner-Goodspeed V, Gallagher J, Gasangwa D, Patxot M, Packiasabapathy S, Mathur P, Eikermann M, Talmor D, Marcantonio ER. Effect of Intravenous Acetaminophen vs Placebo Combined With Propofol or Dexmedetomidine on Postoperative Delirium Among Older Patients Following Cardiac Surgery: The DEXACET Randomized Clinical Trial. JAMA. 2019 Feb 19;321(7):686-696. doi: 10.1001/jama.2019.0234. PMID 30778597
- [Derived] Shankar P, Mueller A, Packiasabapathy S, Gasangwa D, Patxot M, O'Gara B, Shaefi S, Marcantonio ER, Subramaniam B. Dexmedetomidine and intravenous acetaminophen for the prevention of postoperative delirium following cardiac surgery (DEXACET trial): protocol for a prospective randomized controlled trial. Trials. 2018 Jun 22;19(1):326. doi: 10.1186/s13063-018-2718-0. PMID 29929533

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After signing the informed consent, 19 withdrew prior to randomization. (8 patient withdrawals, 8 found ineligible, 1 withdrawn because of inappropriate behavior and emotional lability, 1 withdrawn after entering and receiving intervention in another trial, 1 withdrawn because of inability to complete baseline assessment for same-day admission)
Groups:
- IV Acetaminophen & IV Propofol: 20-100 µg/kg/min IV propofol given for 4-6 hours before the patients are woken up in the ICU
  1g IV acetaminophen every 6 hours for 48 hours during the first 2 days postoperatively
  IV acetaminophen & IV propofol: use of IV tylenol and IV propofol for pain and sedation (respectively)
- IV Acetaminophen & IV Dexmedetomidine: A loading infusion of 0.5 - 1 µg/kg given over 10 minutes will be administered. After the loading infusion, a maintenance infusion of 0.1-1.4 µg/kg/hr will be initiated.
  1 g IV acetaminophen every 6 hours for 48 hours during the first 2 days postoperatively
  IV acetaminophen & IV dexmedetomidine: use of IV tylenol and IV dexmedetomidine for pain and sedation (respectively)
Period: Overall Study
Arm/Group | IV Acetaminophen & IV Propofol | IV Acetaminophen & IV Dexmedetomidine | IV Propofol & Placebo | IV Dexmedetomidine & Placebo
Started | 31 | 30 | 30 | 30
Completed | 31 | 29 (29 Received study drug; 1 withdrew before surgery and after randomization) | 30 | 30
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Acetaminophen-Propofol: Received Intravenous Acetaminophen 6 hourly for 8 doses and intravenous Propofol as sedative until extubation
- Acetaminophen-Dexmedetomidine: Received Intravenous Acetaminophen 6 hourly for 8 doses and intravenous dexmedetomidine as sedative until extubation
- Placebo-Propofol: Received Intravenous Placebo 6 hourly for 8 doses and Intravenous Propofol as a sedative until extubation
- Placebo-Dexmedetomidine: Received Intravenous Placebo 6 hourly for 8 doses and Intravenous Dexmedetomidine as a sedative until extubation
- Total: Total of all reporting groups
Arm/Group | Acetaminophen-Propofol | Acetaminophen-Dexmedetomidine | Placebo-Propofol | Placebo-Dexmedetomidine | Total
Number analyzed (Participants) | 31 | 29 | 30 | 30 | 120
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 70 [66 to 75] | 64 [63 to 72] | 71 [64 to 79] | 69 [63 to 74] | 69 [63 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 4 | 5 | 19
  Male | 24 | 26 | 26 | 25 | 101
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 1 | 4
  Not Hispanic or Latino | 31 | 28 | 28 | 29 | 116
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 1 | 5
  White | 29 | 26 | 28 | 28 | 111
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 31 | 29 | 30 | 30 | 120
Weight [Median (Inter-Quartile Range); unit: kg] | 84.1 [79 to 93.2] | 89.1 [80.4 to 102] | 90 [75.8 to 107] | 87.6 [82 to 102] | 87 [79.15 to 100.15]
Height [Median (Inter-Quartile Range); unit: cms] | 170.2 [167.6 to 173.3] | 173 [167.6 to 180.3] | 175.1 [167.6 to 180] | 172.7 [167.6 to 178] | 172.7 [167.6 to 179]
Body mass index [Median (Inter-Quartile Range); unit: kg/m^2] | 28.5 [26.6 to 32.3] | 29.7 [26.6 to 32.3] | 29.2 [25.9 to 34.3] | 29.4 [27 to 32] | 29.44 [26.53 to 32.69]
Surgical Characteristics- [Number; unit: participants]
  CABG surgery | 19 | 19 | 23 | 18 | 79
  CABG+mitral | 1 | 1 | 0 | 0 | 2
  CABG+aortic | 10 | 8 | 6 | 8 | 32
  Other | 1 | 1 | 1 | 4 | 7
Number of arteries affected [Median (Inter-Quartile Range); unit: arteries] | 3 [2 to 3] | 3 [2 to 4] | 3 [2 to 3] | 3 [2 to 3] | 3 [2 to 3]
Preoperative statin use [Count of Participants; unit: Participants] | 29 | 24 | 27 | 25 | 105
Cross-clamp time [Median (Inter-Quartile Range); unit: minutes] | 78 [66 to 87] | 67 [58 to 84] | 64 [54 to 96] | 73 [60 to 93] | 75 [59 to 93]

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Delirium
Description: Incidence of delirium will be analyzed between patients treated with and without IV acetaminophen, measured from 24 hours post-operation and daily until discharge. Delirium will be defined as an acute change in pre-operative baseline condition with additional features of inattention and either disorganized thinking and altered loss of consciousness, as defined by the Confusion Assessment Method (CAM).
Time Frame: Participants will be followed for the duration of the hospital stay, an average of 5 days
Population: This is a 2 x 2 cross over study.
Measure: Count of Participants; unit: Participants
Groups:
- Acetaminophen and Dexmedetomidine: Patients who received intravenous Acetaminophen for analgesia and dexmedetomidine for sedation
- Acetaminophen and Propofol: Those who received IV acetaminophen for analgesia and Propofol for sedation
- Placebo and Dexmedetomidine: Those who received Placebo for analgesia and dexmedetomidine for sedation
- Placebo and Propofol: Patients who received placebo for analgesia and Propofol for sedation
Arm/Group | Acetaminophen and Dexmedetomidine | Acetaminophen and Propofol | Placebo and Dexmedetomidine | Placebo and Propofol
Number analyzed (Participants) | 29 | 31 | 30 | 30
Participants | 2 | 4 | 8 | 9

2. Secondary Outcome: Duration of Delirium
Description: Duration of delirium will be analyzed, measured from 24 hours post-operation and daily until discharge. Additional measurements will be made at 1 month and 1 year after discharge. Delirium will be defined as an acute change in pre-operative baseline condition with additional features of inattention and either disorganized thinking and altered loss of consciousness, as defined by the Confusion Assessment Method (CAM).
Time Frame: Participants will be followed for the duration of the hospital stay, an average of 6 days, and at 1 month and 1- year following the date of surgery
Population: This is a 2 x 2 cross over study. Therefore, participants were analyzed for primary analgesic use (N=60 in each group)
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Acetaminophen and Dexmedetomidine: Those who received Acetaminophen for analgesia and dexmedetomidine for sedation
- Acetaminophen and Propofol: Those who received acetaminophen for analgesia and propofol for sedation
- Placebo and Propofol: Those who received Placebo for sedation and Propofol for analgesia
Arm/Group | Acetaminophen and Dexmedetomidine | Acetaminophen and Propofol | Placebo and Dexmedetomidine | Placebo and Propofol
Number analyzed (Participants) | 29 | 31 | 30 | 30
days | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 3] | 3 [2 to 3]

3. Secondary Outcome: Severity of Delirium
Description: Severity of delirium will be analyzed, measured from 24 hours post-operation and daily until discharge. The worst severity experienced while in the hospital will be analyzed. Delirium will be defined as an acute change in pre-operative baseline condition with additional features of inattention and either disorganized thinking and altered loss of consciousness, as defined by the Confusion Assessment Method Severity Score (CAM-S, Confusion Assessment Method-Severity). range 0 [best/no delirium] to 19 [worst]; Minimal Clinical Important Difference (MCID) 2 points
Time Frame: Participants will be followed for the duration of the hospital stay, an average of 6 days
Population: This is a 2 x 2 cross over study. Therefore, participants were analyzed for primary analgesic use (N=60 in each group)
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Placebo and Propofol: Those who received placebo for analgesia and propofol for sedation
Arm/Group | Acetaminophen and Dexmedetomidine | Acetaminophen and Propofol | Placebo and Dexmedetomidine | Placebo and Propofol
Number analyzed (Participants) | 29 | 31 | 30 | 30
units on a scale | 10 [9 to 11] | 8 [6 to 10] | 6 [6 to 9] | 9 [8 to 11]

4. Secondary Outcome: Postoperative Opioid Consumption in Morphine Equivalents
Description: Defined by the amount of additional opioid (IV morphine or hydromorphone) and oral acetaminophen medications required in the first 48 hours postoperatively. Values will be converted to morphine equivalents for analysis. Total morphine equivalent is calculated as the sum of (fentanyl dose x 100)+(hydromorphone dose x 4)+morphine dose+(oxycodone dose x 1.5)
Time Frame: Participants will be followed for the first 48 hours postoperatively.
Population: This is a 2 x 2 cross over study.
Measure: Median (Inter-Quartile Range); unit: mcg
Groups:
- Placebo and Propofol: Those who received placebo for analgesia and dexmedetomidine for sedation
Arm/Group | Acetaminophen and Dexmedetomidine | Acetaminophen and Propofol | Placebo and Dexmedetomidine | Placebo and Propofol
Number analyzed (Participants) | 29 | 31 | 30 | 30
mcg | 10050 [5094 to 12530] | 12611 [10026 to 17639] | 11382 [10032 to 18840] | 12616 [10116 to 22590]

5. Secondary Outcome: Montreal Cognitive Assessment (MoCA)
Description: MoCA scores at discharge will be reported in order to assess the occurrence of postoperative cognitive decline. Blinded study staff trained in administering the assessments will collect the data. MoCA is scored on a scale from 0 [worst] to 30 [best]; ǂA MoCA score of 24 would be equivalent to an Mini-Mental State Examination (MMSE) of about 27 or 28. Depending on education and peak intellectual attainment, such a score could be consistent with being either cognitively normal, or having very early mild cognitive impairment. Certainly such a person would be capable of living independently in the community and managing most or all of their affairs.
Time Frame: On the day of discharge, an average of 6 days
Population: This is a 2 x 2 cross over study.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Acetaminophen and Propofol; Placebo and Propofol: Those who received placebo for analgesia and propofol for sedation
Arm/Group | Acetaminophen and Dexmedetomidine | Acetaminophen and Propofol | Placebo and Dexmedetomidine | Placebo and Propofol
Number analyzed (Participants) | 29 | 31 | 30 | 30
score on a scale | 23 [22 to 26] | 24 [22 to 26] | 24 [20 to 26] | 23 [21 to 26]

6. Secondary Outcome: Hospital Length of Stay
Description: Defined by the number of days admitted in the hospital following the completion of surgery.
Time Frame: Measured in days admitted in the hospital, an average of 6 days
Population: This is a 2 x 2 cross over study.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Acetaminophen and Dexmedetomidine | Acetaminophen and Propofol | Placebo and Dexmedetomidine | Placebo and Propofol
Number analyzed (Participants) | 29 | 31 | 30 | 30
days | 8 [6 to 9] | 8 [6 to 11] | 9 [7 to 11] | 8 [6 to 11]

7. Secondary Outcome: ICU Length of Stay
Description: Defined by the number of days admitted in the ICU prior to transfer to the general cardiac surgical floor
Time Frame: Measured in days admitted in the ICU, an average of 2 days
Population: This is a 2 x 2 cross over study.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Acetaminophen and Dexmedetomidine | Acetaminophen and Propofol | Placebo and Dexmedetomidine | Placebo and Propofol
Number analyzed (Participants) | 29 | 31 | 30 | 30
hours | 28.8 [24.9 to 43.5] | 30.3 [25.3 to 52.8] | 49.1 [29 to 92.9] | 29.3 [25.7 to 74.3]

8. Secondary Outcome: Follow up Incidence of Cognitive Dysfunction
Description: The follow up incidence of cognitive dysfunction will be analyzed at 1 month after discharge. T-MoCA is Telephone Montreal Cognitive Assessment Scale (MOCA). The T-MoCA is scored out of 22. The minimum score is 0 (worst) and maximum score is 22 (best). T-MOCA is converted back to 30 (full MOCA) with the help of conversion algorithms to a full MOCA.Example: 19/22 converts back to 30 by performing the following equation: (19×30) ÷ 22. The total converted score is 25.9 or 26/30 which is considered in the normal range.
Time Frame: Patients will be assessed for cognitive dysfunction with T-MOCA at 1 month following the date of surgery
Population: Telephone (T)-MOCA at 1 month. This is a 2 x 2 cross over study.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Acetaminophen and Dexmedetomidine | Acetaminophen and Propofol | Placebo and Dexmedetomidine | Placebo and Propofol
Number analyzed (Participants) | 29 | 31 | 30 | 30
units on a scale | 17 [16 to 20] | 18 [16 to 20] | 19 [17.5 to 21] | 18 [16 to 19.5]

ADVERSE EVENTS:
Time Frame: During hospital stay, an average of 7 days
Description: These were outcomes that are collected by the Society of Thoracic Surgery
Arm/Group | Acetaminophen-Propofol | Acetaminophen-Dexmedetomidine | Placebo-Propofol | Placebo-Dexmedetomidine
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/29 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/29 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 14/31 | 7/29 | 7/30 | 14/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acetaminophen-Propofol (N=31) | Acetaminophen-Dexmedetomidine (N=29) | Placebo-Propofol (N=30) | Placebo-Dexmedetomidine (N=30)
Hypotension (Cardiac disorders) | 14 (14) | 7 (7) | 7 (7) | 14 (14) — Hypotension during the ICU admission
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — ICU bradycardia reported as Heart rate < 60 beats/min

LIMITATIONS AND CAVEATS:
This single center study with restrictive inclusion may place some limitations on generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-29): https://cdn.clinicaltrials.gov/large-docs/65/NCT02546765/Prot_SAP_000.pdf